CLINICAL TRIAL: NCT00988442
Title: A Randomized Trial of Enhanced Nursing Telephone Support to Improve Medication Self-Management and Viral Outcomes of Antiretroviral Therapy-Experienced Patients
Brief Title: Telephone Support to Improve Adherence to Anti-HIV Medications
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was closed to recruitment and follow-up early due to low recruitment.
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ACTG A5251; 1U01AI068636 (NIH); 10632
Record Dates: First submitted 2009-10-01; First posted 2009-10-02 (Estimated); Results first posted 2017-07-17 (Actual); Last update posted 2017-07-17 (Actual); Status verified 2017-04

CONDITIONS: HIV Infections
Keywords: Adherence; Treatment; Adherence Intervention; Telephone Intervention; treatment experienced
MeSH Terms: conditions — HIV Infections; Adherence Interventions | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enhanced nursing telephone support with standard care (Experimental): Participants received enhanced nursing telephone support plus care as usual.
  Interventions: Behavioral: Enhanced nursing telephone support; Behavioral: Standard care
- Standard care (Active Comparator): Participants received care as usual.
  Interventions: Behavioral: Standard care

INTERVENTIONS:
Behavioral: Enhanced nursing telephone support — Weekly phone calls by study nurses for 8 weeks and then calls every 2 weeks for 40 weeks; nurses could schedule more frequent calls at their discretion. Calls provided information, motivational enhancement, problem-solving skills, and affective support.
  Arms: Enhanced nursing telephone support with standard care
Behavioral: Standard care — Usual ACTG site care.

SUMMARY:
This study tested a system of nursing telephone support to determine if it improves adherence to antiretroviral therapy (ART) in at-risk, treatment-experienced people.

DETAILED DESCRIPTION:
Antiretroviral therapy (ART) is only successful in treating HIV when people take all the medications prescribed to them when and how they are instructed. However, a third or more of patients on ART are not able to adhere to their medication regimens. Therefore, making sure that these patients stay healthy involves making sure they are motivated and informed about the importance of adhering to their ART. Nurses can deliver interventions to motivate and inform patients through regularly scheduled phone calls. These calls allow nurses to check in between clinic visits, are convenient to patients, and are cost efficient. This study tested an enhanced telephone support intervention provided by nurses that aimed to improve ART adherence and treatment outcomes.

Follow-up for this study lasted 72 weeks. Participants were randomly assigned to receive either care as usual or the enhanced telephone support intervention plus care as usual. The telephone support intervention involved phone calls made weekly for the first 8 weeks of the study and then every 2 weeks for the next 40 weeks. Nurses made these calls at a time and place participants chose. During the calls, nurses provided information, motivational enhancement, and problem-solving skills.

Study assessments took place at study entry and after 12, 24, 48, and 72 weeks. Assessments measured CD4 cell count, HIV viral load, adherence, and illness events. Adherence was measured through questionnaires and an electronic pill cap.

This study was closed early to both accrual and follow-up due to low recruitment. The study aimed to enroll 296 participants. The actual study accrual at the time of early closing was 59 participants.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in an AIDS Clinical Trials Group (ACTG) treatment study that is an approved A5251 parent or coenrolling partner study ("ACTG parent study participant") or not enrolled in one of the ACTG parent studies, but receiving routine HIV patient care at an institution that was also an ACTG-funded site ("ACTG clinic patient participant").
* Virologic failure on combination antiretroviral therapy (ART), with an HIV-1 genotype conducted on or soon after the failure, within 16 weeks prior to entry. Availability of HIV-1 genotype results at entry.
* History of prior nonadherence to ART during the past year documented either by patient self-report or recorded in the patient's medical record
* Most recent HIV-1 RNA value of at least 200 copies/mL, obtained within 90 days prior to study entry and measured using any FDA-approved test for quantifying HIV-1 RNA
* Initiating or restarting an ART regimen with 2 or more active ARV medications within 3 days after randomization. The regimen must have been selected for the participant prior to the time of randomization for A5251. An active ARV medication was defined as a medication to which the participant was expected to be susceptible based on HIV-1 resistance testing, as specified in the ACTG parent study, or determined by the participant's health care provider per standard of care.

Exclusion Criteria:

* No regular access to a phone. Candidates without phones may have elected to participate by calling the HIV nurse specialists using an 800 number, rather than being called by the HIV nurse specialist.
* Coenrollment in another adherence trial, unless approved by the A5251 study chair
* Current incarceration
* Any condition that, in the opinion of the site investigator, would have compromised the candidate's ability to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy R. Reynolds, PhD, RN, NP, Study Chair — Yale University School of Nursing
Locations (16):
- United States (16):
  - Alabama Therapeutics CRS, Birmingham, Alabama
  - Ucsd, Avrc Crs, San Diego, California
  - Northwestern University CRS (2701), Chicago, Illinois
  - Rush University Medical Center ACTG, Chicago, Illinois
  - Massachusetts General Hospital ACTG CRS, Boston, Massachusetts
  - Bmc Actg Crs (104), Boston, Massachusetts
  - Cooper Univ. Hosp. CRS (31476), Camden, New Jersey
  - New Jersey Medical School-Adult Clinical Research Ctr. CRS, Newark, New Jersey
  - Cornell CRS, New York, New York
  - HIV Prevention & Treatment CRS, New York, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Duke University Medical Center Adult CRS, Durham, North Carolina
  - MetroHealth CRS, Cleveland, Ohio
  - Hospital of the University of Pennsylvania CRS, Philadelphia, Pennsylvania
  - Vanderbilt Therapeutics CRS, Nashville, Tennessee
  - 31443 Trinity Health and Wellness Center CRS, Dallas, Texas

REFERENCES:
- [Background] Reynolds NR, Testa MA, Su M, Chesney MA, Neidig JL, Frank I, Smith S, Ickovics J, Robbins GK; AIDS Clinical Trials Group 731 and 384 Teams. Telephone support to improve antiretroviral medication adherence: a multisite, randomized controlled trial. J Acquir Immune Defic Syndr. 2008 Jan 1;47(1):62-8. doi: 10.1097/QAI.0b013e3181582d54. PMID 17891043
- [Background] Sitta R, Lert F, Gueguen A, Spire B, Dray-Spira R; VESPA group. No variability across centers in adherence and response to HAART in French hospitals: results from the ANRS-EN12-VESPA study. J Acquir Immune Defic Syndr. 2009 Dec;52(5):643-7. doi: 10.1097/QAI.0b013e3181b26eb9. PMID 19668085
- [Background] Zaric GS, Bayoumi AM, Brandeau ML, Owens DK. The cost-effectiveness of counseling strategies to improve adherence to highly active antiretroviral therapy among men who have sex with men. Med Decis Making. 2008 May-Jun;28(3):359-76. doi: 10.1177/0272989X07312714. Epub 2008 Mar 18. PMID 18349433
- [Result] Robbins GK, Cohn SE, Harrison LJ, Smeaton L, Moran L, Rusin D, Dehlinger M, Flynn T, Lammert S, Wu AW, Safren SA, Reynolds NR. Characteristics associated with virologic failure in high-risk HIV-positive participants with prior failure: a post hoc analysis of ACTG 5251. HIV Clin Trials. 2016 Jul;17(4):165-72. doi: 10.1080/15284336.2016.1189754. PMID 27347650

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between April 21, 2011 (first participant enrolled) and October 18, 2012 (last participant enrolled).
Pre-assignment Details: 59 participants were randomized 1:1 to standard care and enhanced nursing telephone support with standard care arms.
Groups:
- Enhanced Nursing Telephone Support With Standard Care: Participants received enhanced nursing telephone support plus care as usual.
  Enhanced nursing telephone support: Weekly phone calls by study nurses for 8 weeks and then calls every 2 weeks for 40 weeks; nurses could schedule more frequent calls at their discretion. Calls provided information, motivational enhancement, problem-solving skills, and affective support.
  Standard care: Care as usual for participants initiating or restarting an ART regimen; this could vary by study site.
- Standard Care: Participants received care as usual.
  Standard care: Care as usual for participants initiating or restarting an ART regimen; this could vary by study site.
Period: Overall Study
Arm/Group | Enhanced Nursing Telephone Support With Standard Care | Standard Care
Started | 30 | 29
Completed | 0 | 1
Not Completed | 30 | 28
Not completed — Death | 1 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Early Study Closure | 29 | 25

BASELINE CHARACTERISTICS:
Population: All participants enrolled in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Enhanced Nursing Telephone Support With Standard Care | Standard Care | Total
Number analyzed (Participants) | 30 | 29 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (12.2) | 46.6 (10.8) | 45.5 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 13 | 23
  Male | 20 | 16 | 36
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Non-Hispanic | 3 | 6 | 9
  Black Non-Hispanic | 23 | 20 | 43
  Hispanic (Regardless of Race) | 4 | 3 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 29 | 59
Intravenous (IV) Drug History [Count of Participants; unit: Participants]
  Never | 26 | 25 | 51
  Previously | 4 | 4 | 8
CD4+ Count [Median (Inter-Quartile Range); unit: cells/mm^3] | 180 [48 to 314] | 157 [82 to 357] | 180 [57 to 333]
HIV-1 RNA [Median (Inter-Quartile Range); unit: log10 copies/mL] | 4.0 [3.1 to 4.9] | 4.5 [3.4 to 4.9] | 4.0 [3.2 to 4.9]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Virologic Suppression
Description: Number of participants with virologic suppression, defined as HIV-1 RNA at less than 200 copies/mL at week 48.
Time Frame: Week 48
Population: All participants enrolled who had Week 48 HIV-1 RNA results available were included in this intent-to-treat-analysis. At the time of early study closure, 14 participants had reached week 48.
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Nursing Telephone Support With Standard Care | Standard Care
Number analyzed (Participants) | 7 | 7
Participants | 4 | 5
Statistical Analysis 1: Comparison: Enhanced Nursing Telephone Support With Standard Care vs Standard Care; A Fisher's exact test was used to compare the proportion of participants with virologic suppression, defined as HIV-1 RNA less than 200 copies/mL at week 48 between the standard of care and standard of care + enhanced telephone support groups; Test type: Superiority or Other; p = 1.000, Fisher Exact — Two-sided 5% significance level

2. Secondary Outcome: Number of Participants With Premature Antiretroviral Therapy (ART) Regimen Discontinuation
Description: Number of premature ART regimen discontinuations, defined as the first substitution, subtraction, or addition of one or more ARVs made to the initial study regimen.
Time Frame: From study entry to Week 72
Population: All participants with available ART data.
Measure: Number; unit: participants
Arm/Group | Enhanced Nursing Telephone Support With Standard Care | Standard Care
Number analyzed (Participants) | 30 | 28
participants | 4 | 7

3. Secondary Outcome: Change in CD4 Cell Count at Week 12
Description: Change in CD4 cell count from baseline at week 12, calculated as Week 12 CD4 minus baseline CD4.
Time Frame: Baseline and Week 12
Population: Due to early study closure, only 44 participants had week 12 CD4 observations to be included in this analysis.
Measure: Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | Enhanced Nursing Telephone Support With Standard Care | Standard Care
Number analyzed (Participants) | 22 | 22
cells/mm^3 | 11 [-12 to 35] | 27 [-12 to 67]

4. Secondary Outcome: Change in CD4 Cell Count at Week 24
Description: Change in CD4 cell count from baseline at Week 24, calculated as Week 24 CD4 minus baseline CD4.
Time Frame: Baseline and Week 24
Population: Due to early study closure, only 42 participants had week 24 CD4 observations to be included in this analysis.
Measure: Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | Enhanced Nursing Telephone Support With Standard Care | Standard Care
Number analyzed (Participants) | 21 | 21
cells/mm^3 | 37 [-3 to 77] | 9 [-32 to 51]

5. Secondary Outcome: Change in CD4 Cell Count at Week 48
Description: Change in CD4 cell count from baseline at Week 48, calculated as Week 48 CD4 minus baseline CD4.
Time Frame: Baseline and Week 48
Population: Only 16 participants had week 48 CD4 observations to be included in this analysis.
Measure: Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | Enhanced Nursing Telephone Support With Standard Care | Standard Care
Number analyzed (Participants) | 8 | 8
cells/mm^3 | 63 [-64 to 189] | 80 [4 to 156]

6. Secondary Outcome: Confirmed Virologic Failure
Description: Number of participants with confirmed virologic failure. Virologic failure is defined as confirmed HIV-1 RNA ≥200 copies/mL at or after the week 24 HIV-1 RNA evaluation (obtained at least 20 weeks after the date of randomization).
Time Frame: Week 24 through Week 72
Population: The analysis population was all participants randomized to a treatment arm in this trial.
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Nursing Telephone Support With Standard Care | Standard Care
Number analyzed (Participants) | 30 | 29
Participants
  Virologic Failure | 8 | 7
  Virologic Non-failure | 6 | 6
  Insufficient Follow Up | 16 | 16

7. Secondary Outcome: Cost of the Adherence Telephone Interventions
Description: This outcome was planned to be analyzed if the intervention was found to be successful. However, the intervention was not determined to be successful.
Time Frame: Week 48
Population: This outcome was not analyzed, since the intervention was not determined to be successful.
Arm/Group | Enhanced Nursing Telephone Support With Standard Care | Standard Care
Number analyzed (Participants) | 0 | 0
Value | 0 | 0

8. Secondary Outcome: Number of Participants With Illness Events or Mortality
Description: Number of participants who had acute illnesses and mortality during follow-up. The categories of illness events and mortality are not mutually exclusive.
Time Frame: Measured from entry to Week 72 or premature study discontinuation
Population: Due to early study closure, only 59 participants were accrued and followed on study.
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Nursing Telephone Support With Standard Care | Standard Care
Number analyzed (Participants) | 30 | 29
Participants
  Fungal infections | 2 | 5
  Bacterial/Mycobacterial infections | 5 | 3
  Viral infections | 1 | 4
  Neoplastic diseases | 1 | 1
  Cardiovascular diseases | 5 | 2
  Other Disease - General Diagnoses | 6 | 4
  Other Disease - Metabolic/Endocrine | 3 | 0
  Other Disease - Pulmonary | 4 | 2
  Other Disease - Gastrointestinal | 5 | 4
  Other Disease - Genitourinary | 1 | 2
  Other Disease - Neuropsychiatric | 4 | 2
  Other Disease - Musculoskeletal | 1 | 0
  Other Disease - Dermatologic | 3 | 0
  Other Disease - STD | 0 | 1
  Other HIV Associated Diseases | 0 | 2
  Deaths | 1 | 2

9. Secondary Outcome: Number of Participants With Virological Suppression
Description: Number of participants with virological suppression, defined as HIV-1 RNA less than 200 copies/mL.
Time Frame: Measured from entry to Week 72 or premature study discontinuation
Population: All participants with scheduled post baseline HIV-1 RNA measurements.
Measure: Number; unit: participants
Arm/Group | Enhanced Nursing Telephone Support With Standard Care | Standard Care
Number analyzed (Participants) | 26 | 27
participants | 14 | 15

10. Secondary Outcome: Number of Participants Who Received Last Telephone Call if Prior to the End of Defined Intervention Period
Description: Number of participants whose last telephone call received occurred prior to the end of the defined intervention period.
Time Frame: Measured from entry to Week 72 or premature study discontinuation
Population: Only participants in the telephone support group were analyzed.
Measure: Number; unit: participants
Arm/Group | Enhanced Nursing Telephone Support With Standard Care | Standard Care
Number analyzed (Participants) | 30 | 0
participants | 21 |

11. Secondary Outcome: Intervention Dosage Score for Enhanced Nursing Telephone Support (Total Percentage of Scheduled Calls Successfully Delivered)
Description: Intervention dosage score for enhanced nursing telephone support. This is the total percentage of scheduled calls successfully delivered.
Time Frame: Measured at Week 12
Population: Only participants in the telephone support group were analyzed.
Measure: Mean (Standard Deviation); unit: percent of scheduled calls delivered
Arm/Group | Enhanced Nursing Telephone Support With Standard Care | Standard Care
Number analyzed (Participants) | 30 | 0
percent of scheduled calls delivered | 34.6 (34.3) |

12. Secondary Outcome: Intervention Dosage Score for Enhanced Nursing Telephone Support (Total Amount of Time Spent in Calls)
Description: Intervention dosage score for enhanced nursing telephone support. This is the total amount of time spent in calls overall.
Time Frame: Week 12
Population: Only participants in the telephone support group were analyzed.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Enhanced Nursing Telephone Support With Standard Care | Standard Care
Number analyzed (Participants) | 30 | 0
minutes | 19 [0 to 39] |

13. Secondary Outcome: Number of Participants With Virologic Suppression, Defined as HIV-1 RNA Less Than 200 Copies/mL at Week 12
Description: Number of participants with virologic suppression, defined as HIV-1 RNA less than 200 copies/mL, at week 12.
Time Frame: Week 12
Population: Due to early study closure, only the 43 participants who reached week 12 with available virologic data were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Nursing Telephone Support With Standard Care | Standard Care
Number analyzed (Participants) | 21 | 22
Participants | 10 | 12

14. Secondary Outcome: Number of Participants With Virologic Suppression, Defined as HIV-1 RNA Less Than 200 Copies/mL at Week 24.
Description: Number of participants with virologic suppression, defined as HIV-1 RNA less than 200 copies/mL, at week 24.
Time Frame: Week 24
Population: Due to early study closure, only the 41 participants who reached week 24 with available data were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Nursing Telephone Support With Standard Care | Standard Care
Number analyzed (Participants) | 22 | 19
Participants | 10 | 7

15. Secondary Outcome: Number of Participants With Virologic Suppression, Defined as HIV-1 RNA Less Than 1,000 Copies/mL at Week 12
Description: Number of participants with virologic suppression, defined as HIV-1 RNA less than 1,000 copies/mL, at week 12.
Time Frame: Week 12
Population: Due to early study closure, only the 43 participants who reached week 12 with available data were included in this analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Standard Care: Participants received care as usual.
  Standard care: Care as usual for participants initiating or restarting an ART regimen; this may vary by study site.
Arm/Group | Enhanced Nursing Telephone Support With Standard Care | Standard Care
Number analyzed (Participants) | 21 | 22
Participants | 12 | 13

16. Secondary Outcome: Number of Participants With Virologic Suppression, Defined as HIV-1 RNA Less Than 1,000 Copies/mL at Week 24
Description: Number of participants with virologic suppression, defined as HIV-1 RNA less than 1,000 copies/mL, at week 24.
Time Frame: Week 24
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Nursing Telephone Support With Standard Care | Standard Care
Number analyzed (Participants) | 22 | 19
Participants | 11 | 8

17. Secondary Outcome: Number of Participants With Virologic Suppression, Defined as HIV-1 RNA Less Than 1,000 Copies/mL at Week 48
Description: Number of participants with virologic suppression, defined as HIV-1 RNA less than 1,000 copies/mL, at week 48.
Time Frame: Measured at Week 48
Population: Due to early study closure, only the 14 participants that reached week 48 with available data were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Nursing Telephone Support With Standard Care | Standard Care
Number analyzed (Participants) | 7 | 7
Participants | 5 | 5

18. Secondary Outcome: Antiretroviral (ARV) Medication Adherence at Week 12 Using ACTG Adherence Questionnaire
Description: ARV medication adherence at week 12, as measured by the ACTG adherence questionnaire index. This questionnaire index is on a 0-100 scale, with higher scores indicating higher adherence.
Time Frame: Week 12
Population: Due to early study closure, only 30 participants had complete adherence data for this outcome.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Enhanced Nursing Telephone Support With Standard Care | Standard Care
Number analyzed (Participants) | 16 | 14
units on a scale | 97 [79 to 99] | 93 [83 to 98]

19. Secondary Outcome: Antiretroviral (ARV) Medication Adherence at Week 24 Using ACTG Adherence Questionnaire
Description: ARV medication adherence at week 24, as measured by the ACTG adherence questionnaire index. The ACTG adherence questionnaire index is on a 0-100 scale where higher scores indicate better adherence.
Time Frame: Week 24
Population: Due to early study closure, 31 participants had complete adherence data for this outcome.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Enhanced Nursing Telephone Support With Standard Care | Standard Care
Number analyzed (Participants) | 15 | 16
units on a scale | 91 [52 to 99] | 95 [67 to 98]

20. Secondary Outcome: Antiretroviral (ARV) Medication Adherence at Week 12 Using Four Day Recall
Description: ARV medication adherence at week 12, as measured by four day recall, i.e. "Missed doses in last 4 days".
Time Frame: Week 12
Population: Due to early study closure, only 42 participants had adherence data at week 12 for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Nursing Telephone Support With Standard Care | Standard Care
Number analyzed (Participants) | 23 | 19
Participants
  Missed Doses: 0 | 17 | 16
  Missed Doses: 1-2 | 0 | 1
  Missed Doses: 3-4 | 3 | 1
  Missed Doses: 5+ | 3 | 1

21. Secondary Outcome: Antiretroviral (ARV) Medication Adherence at Week 24 Using Four Day Recall
Description: ARV medication adherence, as measured by four day recall, i.e. "Missed doses in last 4 days".
Time Frame: Week 24
Population: Due to early study closure, only 39 participants had adherence data at week 24.
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Nursing Telephone Support With Standard Care | Standard Care
Number analyzed (Participants) | 21 | 18
Participants
  Missed Doses: 0 | 12 | 11
  Missed Doses: 1-2 | 1 | 1
  Missed Doses: 3-4 | 2 | 3
  Missed Doses: 5+ | 6 | 3

22. Secondary Outcome: Antiretroviral (ARV) Medication Adherence at Week 12 Using Visual Analog Scale
Description: ARV medication adherence at week 12, as measured by the visual analog scale. The visual analog scale is a 0-100% scale that measures the percentage of HIV medication taken in the past month.
Time Frame: Week 12
Population: Due to early study closure, only 44 participants had adherence data available at week 12 for this outcome.
Measure: Median (Inter-Quartile Range); unit: percentage of HIV meds taken last month
Arm/Group | Enhanced Nursing Telephone Support With Standard Care | Standard Care
Number analyzed (Participants) | 23 | 21
percentage of HIV meds taken last month | 95 [55 to 100] | 95 [85 to 100]

23. Secondary Outcome: Antiretroviral (ARV) Medication Adherence at Week 24 Using Visual Analog Scale
Description: ARV medication adherence at Week 24, as measured by the visual analog scale. The visual analog scale is a 0-100% scale that measures the percentage of HIV medication taken in the past month.
Time Frame: Week 24
Population: Due to early study closure, only 40 participants had adherence data available at week 24 for this outcome.
Measure: Median (Inter-Quartile Range); unit: percentage of HIV meds taken last month
Arm/Group | Enhanced Nursing Telephone Support With Standard Care | Standard Care
Number analyzed (Participants) | 21 | 19
percentage of HIV meds taken last month | 95 [60 to 100] | 95 [70 to 100]

24. Secondary Outcome: Quality of Life Measured by Euro-QoL - Mobility
Description: Quality of life measured by Euro-QoL - Question 1: Mobility.
Time Frame: Week 24
Population: Available data for participants that reached week 24 are summarized.
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Nursing Telephone Support With Standard Care | Standard Care
Number analyzed (Participants) | 22 | 19
Participants
  No problems walking | 18 | 11
  Some problems walking | 4 | 8

25. Secondary Outcome: Quality of Life Measured by Euro-QoL - Self-Care
Description: Quality of Life Measured by Euro-QoL - Question 2: Self-Care.
Time Frame: Week 24
Population: All available data from participants that reached week 24 are summarized.
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Nursing Telephone Support With Standard Care | Standard Care
Number analyzed (Participants) | 22 | 19
Participants
  No problems with self-care | 21 | 18
  Some problems washing or dressing | 1 | 1

26. Secondary Outcome: Quality of Life Measured by Euro-QoL - Usual Activities
Description: Quality of Life Measured by Euro-QoL - Question 3: Usual activities.
Time Frame: Week 24
Population: All available data from participants that reached week 24 are summarized.
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Nursing Telephone Support With Standard Care | Standard Care
Number analyzed (Participants) | 22 | 19
Participants
  No problems performing usual activities | 20 | 16
  Some probs performing usual activities | 1 | 3
  Unable to perform usual activities | 1 | 0

27. Secondary Outcome: Quality of Life Measured by Euro-QoL - Pain/Discomfort
Description: Quality of Life Measured by Euro-QoL - Question 4: Pain/Discomfort.
Time Frame: Week 24
Population: Available data from participants who reached week 24 are summarized.
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Nursing Telephone Support With Standard Care | Standard Care
Number analyzed (Participants) | 22 | 19
Participants
  No pain or discomfort | 14 | 9
  Moderate pain or discomfort | 6 | 5
  Extreme pain or discomfort | 2 | 5

28. Secondary Outcome: Quality of Life Measured by Euro-QoL - Anxiety/Depression
Description: Quality of Life Measured by Euro-QoL - Question 5: Anxiety/Depression.
Time Frame: Week 24
Population: Available data from participants who made it to week 24 are summarized.
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Nursing Telephone Support With Standard Care | Standard Care
Number analyzed (Participants) | 22 | 19
Participants
  Not anxious or depressed | 17 | 10
  Moderately anxious or depressed | 3 | 8
  Extremely anxious or depressed | 2 | 1

ADVERSE EVENTS:
Time Frame: Measured from entry to Week 72 or premature study discontinuation
Description: No adverse event data other than number of deaths were collected in this study.
Groups:
- Enhanced Nursing Telephone Support With Standard Care: Participants will receive enhanced nursing telephone support plus care as usual.
  Enhanced nursing telephone support: Weekly phone calls by study nurses for 8 weeks and then calls every 2 weeks for 40 weeks; nurses may schedule more frequent calls at their discretion. Calls will provide information, motivational enhancement, problem-solving skills, and affective support.
  Standard care: Care as usual for participants starting a new ART regimen; this may vary by study site.
- Standard Care: Participants will receive care as usual.
  Standard care: Care as usual for participants starting a new ART regimen; this may vary by study site.
Arm/Group | Enhanced Nursing Telephone Support With Standard Care | Standard Care
All-Cause Mortality (participants affected / at risk) | 1/30 | 2/29
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
This study was closed to recruitment and follow-up early due to slow enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No